CLINICAL TRIAL: NCT02706626
Title: Phase 2 Trial of Brigatinib After Treatment With Next-Generation ALK Inhibitors in Refractory ALK Rearranged Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Trial of Brigatinib After Treatment With Next-Generation ALK Inhibitors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not meet enrollment objectives.
Sponsor: Criterium, Inc. (Industry)
Collaborators: University of Colorado, Denver (Other); Duke University (Other); Takeda (Industry); Vanderbilt University (Other); University of Texas Southwestern Medical Center (Other); University of Pittsburgh (Other); Ohio State University (Other); Georgetown University (Other); Academic Thoracic Oncology Medical Investigators Consortium (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARI-AT-002
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — brigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Disease progression after next generation ALK TKI (Experimental): Brigatinib until progressive disease, unacceptable toxicity, withdrawal of consent. Patients enrolled regardless the number of lines of therapy
  Interventions: Drug: brigatinib
- Cohort B: Disease progression after alectinib as first-line therapy (Experimental): Brigatinib until progressive disease, unacceptable toxicity, withdrawal of consent. Patients enrolled after first-line alectinib
  Interventions: Drug: brigatinib
- Cohort C: Disease progression after brigatinib (Experimental): Brigatinib at 240 mg daily until progressive disease, unacceptable toxicity, withdrawal of consent. Patients enrolled after treatment on brigatinib at the standard dose brigatinib
  Interventions: Drug: brigatinib

INTERVENTIONS:
Drug: brigatinib — Single arm phase 2 trial to investigate the clinical activity in patients with advanced non-small cell lung cancer
  Other Names: AP26113

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of this investigational drug, brigatinib (AP261136) in patients with advanced non-small cell lung cancer Non-small cell lung cancer (NSCLC) who have had first-line treatment for their cancer and it still got worse, even after, or while taking drugs called ALK inhibitors, or anti-cancer drugs that act on tumors. Some examples of these anti-cancer drugs are: KEYTRUDA® or ALECENSA®).

DETAILED DESCRIPTION:
A significant population of Anaplastic Lymphoma Kinase (ALK) plus Non-small cell lung cancer patients exist that have progressed on or who were intolerant of second generation anaplastic lymphoma kinase inhibitor (e.g. ceritinib or alectinib). Brigatinib has demonstrated activity in patients who have progressed on crizotinib, but the activity of brigatinib in patients who have progressed on ceritinib, alectinib, or other second generation anaplastic lymphoma kinase inhibitors is unknown. Based on the preclinical data. 3, , brigatinib has activity against known secondary anaplastic lymphoma kinase mutations suggesting it may retain activity after second-generation anaplastic lymphoma kinase inhibitors.

Patients enrolled in ARI-AT-002 must have previously received a second generation Anaplastic lymphoma kinase inhibitor other than brigatinib. We have chosen 20% as a clinically meaningful response rate that would justify further study of brigatinib in previously treated anaplastic lymphoma kinase plus disease.

ELIGIBILITY:
Inclusion Criteria:

Locally advanced or metastatic NSCLC that has been cytologically or histologically confirmed

ALK rearrangement based on FDA approved test (e.g. Vysis breakapart FISH or IHC using Ventana)

ECOG PS ≤2

Age of ≥ 18 years

Brain lesions may be used as target lesions if progressing, ≥10mm in longest diameter and if they were not previously treated with any of the following:

* Whole brain radiation therapy (WBRT) within 3 months
* Stereotactic radiosurgery (SRS)
* Surgical resection Availability of core biopsy of progressive lesion taken within 60 days prior to D1 of treatment under study therapy or willing to undergo tumor biopsy: NOTE:. All subjects must consent to provide tumor blocks or slides.
* If archival tissue is not available and biopsies to obtain fresh tumor tissue cannot be performed with minimal risk to the subject, subjects may be permitted to enroll on the study with prior approval of the Study PI.
* In the situation the patient undergoes biopsy within 60 days prior to D1. and there is insufficient tumor tissue subjects for the correlative science part of the protocol patient will be permitted to enroll on the study with prior approval of the study PI
* In the situation the patient undergoes molecular testing or next-generation sequencing as part of standard care there must be sufficient tumor sample available for participation in the study (i.e. a next generation sequencing report is not sufficient for enrollment)

Recovered from toxicities related to prior anticancer treatment to ≤Grade 2 or baseline with the exception of alopecia

Have normal QT interval on ECG evaluation QT corrected Fridericia (QTcF) of ≤ 450 ms in males or ≤ 470 ms in females

Adequate organ function defined as:

Absolute neutrophil count (ANC) ≥1500/µL Platelets ≥75,000/µL Hemoglobin≥ 10g/dL AST /ALT ≤ 2.5 x upper limit of normal (ULN); ≤ 5 x ULN if liver metastasis Total serum bilirubin ≤ 1.5 x ULN Serum creatinine ≤ 1.5 x UNL Serum amylase ≤ 1.5 x UNL

At least 1 measurable lesion per RECIST version 1.1

Negative serum pregnancy test within 7 days of D1 of treatment in women of child bearing potential (WOCBP)

If fertile, willing to use highly effective form of contraception (defined as a combination of at least two of the following methods: condom or other barrier methods, oral contraceptives, implantable contraceptives, intrauterine devices) during the dosing period and for at least 4 months after

Ability to provide signed informed consent and willing and able to comply with all study requirements

Inclusion criteria for cohort assignment:

Cohort A: Progressive disease on any next generation ALK inhibitor except first line alectinib or brigatinib (any line)

Cohort B: Progressive disease on first-line therapy with alectinib, and no other ALK inhibitors

Cohort C: Previous treatment brigatinib at 180 mg daily for ≥4 weeks without > grade 2 drug-related toxicities and with radiographic evidence of progressive disease and no intervening systemic therapies such as chemotherapy, immunotherapy or another ALK inhibitor (radiation therapy allowed as intervening therapy). Patients who are treated on cohorts A and B will be allowed to enroll in cohort C if the meet the inclusion and exclusion criteria

Exclusion Criteria for cohorts A, B, and C:

Patients meeting any of the following exclusion criteria will not be able to participate in this study:

History or the presence of pulmonary interstitial disease, drug-related or immune-related pneumonitis, or radiation pneumonitis requiring medical management within 6 months of trial enrollment

Prior treatment with brigatinib for cohorts A and B

History of or active significant gastrointestinal (GI) bleeding within 3 months

Malabsorption syndrome or other GI illness that could affect oral absorption of the study drug

Received cytotoxic chemotherapy, investigational agents or radiation within 7 days prior to D1 of study treatment

Received prior ALK TKI therapy within 7 days prior to D1 of treatment under study drug. 7 day wash out period is required after prior ALK inhibitor treatment.

Have significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

* Myocardial infarction (MI) within 6 months of trial enrollment
* Unstable angina within 6 months of trial enrollment
* Congestive heart failure (CHF) with 6 months prior to trial enrollment
* Any history of ventricular arrhythmia
* Cerebrovascular accident or transient ischemic attack within 6 months of D1 of study treatment
* Clinically significant atrial arrhythmia or severe baseline bradycardia defined as resting heart rate < 60 beat per minute
* Uncontrolled hypertension defined as baseline SBP> 160 and DBP > 100 on 3 separate clinic visits or past history of hypertensive urgency, emergency or encephalopathy

Have been diagnosed with another primary malignancy within the past 3 years (except for adequately treated non-melanoma skin cancer, cervical cancer in situ, or prostate cancer, which are allowed within 3 years)

Have symptomatic CNS metastases which require an increasing dose of corticosteroids within the last 2 weeks to remain asymptomatic.

Have active infection requiring intravenous antibiotics

Pregnant or breastfeeding

Have any condition or illness that, in the opinion of the investigator, would compromise patient safety or interfere with evaluation of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Stinchcombe, MD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - University Of Colorado, Denver, Colorado
  - Duke University, Durham, North Carolina
  - Vanderbilt Unversity Medical Center, Nashville, Tennessee
  - University of Texas, Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stinchcombe TE, Doebele RC, Wang X, Gerber DE, Horn L, Camidge DR. Preliminary Clinical and Molecular Analysis Results From a Single-Arm Phase 2 Trial of Brigatinib in Patients With Disease Progression After Next-Generation ALK Tyrosine Kinase Inhibitors in Advanced ALK+ NSCLC. J Thorac Oncol. 2021 Jan;16(1):156-161. doi: 10.1016/j.jtho.2020.09.018. Epub 2020 Oct 8. PMID 33039599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study closed before total enrollment expectations were met.
Pre-assignment Details: The clinical trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results. Patient were enrolled in the trial and were assigned based on previous treatment
Groups:
- Arm A: Brigatinib After Next Generation ALK TKI: Patients with disease progression after next generation ALK TKI
- Arm B: Patients Disease Progression After First-line Alectinib: Patients were required to have disease progression after first-line alectinib
- Arm C: Brigatinib 240 mg for Patients With Disease Progression on Brigatinib: Patients had disease progression on standard dose brigatinib and experience disease progression
Period: Overall Study
Arm/Group | Arm A: Brigatinib After Next Generation ALK TKI | Arm B: Patients Disease Progression After First-line Alectinib | Arm C: Brigatinib 240 mg for Patients With Disease Progression on Brigatinib
Started | 27 | 4 | 1 (3 subjects from cohort A transitioned to cohort C, total unique subjects = 32)
Completed | 27 | 4 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients were enrolled and assigned to a cohort based on previous treatment. Cohort A enrolled patients with disease progression on a next generation ALK TKI regardless of the number of lines of therapy. Cohort B enrolled patients who had received first line alectinib. Cohort C enrolled patients with disease progression on standard dose brigatinib and who tolerated the therapy
Groups:
- Cohort A: Disease Progression After Next Generation ALK TK: Patients could enroll in this cohort after a next generation ALK TKI (regardless of the number of previous therapies)
- Cohort B: Disease Progression After Alectinib as First-line Therapy: Patients could enroll in this cohort after first-line alectinib
- Arm C: Brigatinib 240 mg for Patients With Disease Progression on Brigatinib: Patients who tolerated standard dose brigatinib and had disease progression could enroll in this cohort
- Total: Total of all reporting groups
Arm/Group | Cohort A: Disease Progression After Next Generation ALK TK | Cohort B: Disease Progression After Alectinib as First-line Therapy | Arm C: Brigatinib 240 mg for Patients With Disease Progression on Brigatinib | Total
Number analyzed (Participants) | 27 | 4 | 1 | 32
Age, Customized [Median (Full Range); unit: years]
  Median Age | 57 [32 to 74] | 43 [39 to 51] | 76 [56 to 76] | 56 [32 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 1 | 0 | 12
  Male | 16 | 3 | 1 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23 | 3 | 1 | 27
  African American | 1 | 0 | 0 | 1
  Latino or Hispanic | 1 | 0 | 0 | 1
  Asian | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: An assessment of the response using RECIST 1.1 per investigator. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.". The enrollment in the clinical trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results
Time Frame: Through study completion (average 42 months)
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Brigatinib After Next Generation ALK TKI Regardless of Number of Therapies: Patients with disease progression after next generation ALK TKI as first or second-line therapy, regardless of number of therapies
- Arm B: Brigatinib After First-line Therapy With Alectinib: Patient were treated with first-line alectinib and had disease progression
- Arm C: Brigatinib 240 mg in Patient With Disease Progression on Brigatinib 180 mg Daily: Patients had disease control on brigatinib and then experience disease progression and did not have severe toxicities related brigatinib
Arm/Group | Arm A: Brigatinib After Next Generation ALK TKI Regardless of Number of Therapies | Arm B: Brigatinib After First-line Therapy With Alectinib | Arm C: Brigatinib 240 mg in Patient With Disease Progression on Brigatinib 180 mg Daily
Number analyzed (Participants) | 27 | 4 | 4
Participants | 9 | 1 | 0

ADVERSE EVENTS:
Time Frame: Patients were followed until disease progression or unacceptable toxicity or withdrawal of consent, on average 1 year
Groups:
- Arm A: Brigatinib After Next Generation ALK TKI: Patients had disease progression on any next generation ALK TKI (regardless of the number of lines of therapy)
- Arm B: Brigatinib After First-line Alectinib: Patients had disease progression on first line alectinib, and not additional therapies were allowed
- Arm C: Brigatinib 240 mg in Patients With Disease Progression on Brigatinb: Patients had disease progression on standard dose brigatinib who tolerated standard dose brigatinib
Arm/Group | Arm A: Brigatinib After Next Generation ALK TKI | Arm B: Brigatinib After First-line Alectinib | Arm C: Brigatinib 240 mg in Patients With Disease Progression on Brigatinb
All-Cause Mortality (participants affected / at risk) | 10/27 | 1/4 | 1/4
Serious Adverse Events (participants affected / at risk) | 8/27 | 2/4 | 2/4
Other Adverse Events (participants affected / at risk) | 11/27 | 1/4 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Brigatinib After Next Generation ALK TKI (N=27) | Arm B: Brigatinib After First-line Alectinib (N=4) | Arm C: Brigatinib 240 mg in Patients With Disease Progression on Brigatinb (N=4)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis, pleural effusion,hemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2)
Increased CPK (Investigations) | 2 (2) | 0 (0) | 0 (0)
Muscle or bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Brigatinib After Next Generation ALK TKI (N=27) | Arm B: Brigatinib After First-line Alectinib (N=4) | Arm C: Brigatinib 240 mg in Patients With Disease Progression on Brigatinb (N=4)
Lab abnormalities (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anrorexia fatigue, (General disorders) | 1 (1) | 0 (0) | 0 (0)
Headaches, dizzimes (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cough, shortness of breath, dsypnea, upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
Increased creatinine (Renal and urinary disorders) | 4 (4) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated for slow accrual. The enrollment in the clinical trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT02706626/Prot_SAP_000.pdf
  • Informed Consent Form: Main ICF (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT02706626/ICF_001.pdf
  • Informed Consent Form: Addendum to ICF (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT02706626/ICF_002.pdf